CLINICAL TRIAL: NCT04709718
Title: Surgical Management of Giant Hepatic Hemangioma: a 10-year Single Center Experience
Brief Title: Surgical Management of Giant Hepatic Hemangioma
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Collaborators: Sahloul Hospital of Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, clinical professor, Université de Sousse
Other Study IDs: U23464
Record Dates: First submitted 2021-01-01; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Liver Angioma
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- churgery of geant liver hemangioma
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: hepatectomy — liver resection taking over the liver hemangioma

SUMMARY:
Hepatic hemangiomas are the commonest benign mesenchymal lesions of the liver. Most of these lesions are asymptomatic. Giant hepatic hemangiomas (GHH) (> 10 cm) are often symptomatic and require surgical intervention. This study aimed to describe the clinical findings, risk factors, diagnostic approach and management of GHH.

DETAILED DESCRIPTION:
Hepatic hemangiomas are the most common benign tumors of the liver with the incidence of 0.4 to 20% . They are most often discovered incidentally on imaging studies. Typical hemangiomas usually do not increase in size over time and therefore are unlikely to cause symptoms. Giant hepatic hemangiomas (GHH) are defined as hemangiomas larger than 5 cm . They are usually responsible for overt clinical symptoms and complications consisting, most often, of upper abdominal pain, hemorrhage, biliary compression, or a consumptive coagulopathy that may require prompt surgical intervention or other treatments . Management of liver hemangiomas ranges from close observation to surgery depending upon the site, size and symptoms .

It is widely accepted that intervention is indicated only for symptomatic hemangiomas. Surgical resection is indicated in patients with abdominal complaints or complications, or when diagnosis remains inconclusive. The ideal surgical treatment for GHH is still controversial. Enucleation is the preferred surgical method based on the existing literature. In this study, we report our 17-year experience of clinical management of GHH.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of geant liver hamangioma.

Exclusion Criteria:

* Radiological diagnosis of liver hemangioma less than 10cm.

Ages: 15 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patient with symptomatic geant liver hemangioma
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
number of patient getting good result after surgery | 1 year
  patient asymptomatic after surgery or not

CONTACTS AND LOCATIONS:
Overall Officials: waad farhat, doctor, Study Director — university of sousse

IPD SHARING:
Plan to Share IPD: Undecided